CLINICAL TRIAL: NCT02263677
Title: Pilot Project Evaluation of the DPP-4 Inhibitor Sitagliptin in the Treatment of Non-Alcoholic Fatty Liver Disease Using MRI
Brief Title: Evaluation of the DPP-4 Inhibitor Sitagliptin in the Treatment of Non-Alcoholic Fatty Liver Disease Using MRI
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Technical difficulties have caused this study to be terminated
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MERCK-9938
Record Dates: First submitted 2014-10-01; First posted 2014-10-13 (Estimated); Last update posted 2016-10-05 (Estimated); Status verified 2016-10

CONDITIONS: Type 2 Diabetes; Non-alcoholic Fatty Liver Disease
Keywords: diabetes; fatty liver
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Non-alcoholic Fatty Liver Disease; Diabetes Mellitus; Fatty Liver | interventions — Sitagliptin Phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sitagliptin (Experimental): 60 day supply of 100mg Sitagliptin
  Interventions: Drug: Sitagliptin

INTERVENTIONS:
Drug: Sitagliptin — 60 day supply of 100mg Sitagliptin. The investigators will use an MRS (a non invasive method using magnets) to evaluate liver fat before and after subjects take a diabetes medication. The investigators will also collect a small amount of blood to measure liver, kidney and hormone functions. This will be done 4 times. Also, at the time of the subject gets their first dose of medication they will have a DEXA (low exposure x-ray often used in clinical practice to measure bone density and body composition).
  Other Names: Januvia

SUMMARY:
Participants will be persons with type 2 diabetes who are likely to have fatty liver disease. The investigators think that this medication will reduce fatty liver.

The investigators will use an MRS (a non invasive method using magnets) to evaluate liver fat before and after subjects take a diabetes medication. The investigators will also collect a small amount of blood to measure liver, kidney and hormone functions. This will be done 4 times. Also, at the time of the subject gets their first dose of medication they will have a DEXA (low exposure x-ray often used in clinical practice to measure bone density and body composition).

The goal of all of these studies is to determine whether the study drug lowers liver fat.

DETAILED DESCRIPTION:
Non-alcoholic fatty liver disease (NAFLD) and its progression to non-alcoholic steatohepatitis (NASH) and finally cirrhosis is rapidly becoming the leading cause of liver injury and end stage liver disease, particularly in industrialized countries. Though several pharmacologic agents (i.e. metformin, pioglitazone and others) have been suggested to have benefit in reducing the progression of this disease, none is approved for use.

The causes of NAFLD and NASH are unknown, though visceral obesity, metabolic syndrome and type 2 diabetes are recognized co-existent risk factors. Recent evidence has linked NAFLD to elevated dipeptidyl peptidase-4 (DPP-4). DPP-4 levels in the plasma and livers of persons with NAFLD are elevated and correlate with elevations in liver enzymes, though not with markers of insulin resistance alone.

It has been proposed that increased DPP-4 activity in combination with decreased PPAR signaling stimulates the inflammatory response that leads to liver fibrosis in the transition of NASH to cirrhosis. Debate exists as to whether the effect of DPP-4 in the liver is via its effect on the intestinal hormones or its direct effects on liver tissue. Indeed some studies have found reductions in liver fat with administration of GLP-1 agonists in animal models of obesity.

ELIGIBILITY:
Inclusion Criteria:

1. Type 2 diabetes mellitus with hemoglobin A1c above 6.5%.
2. Waist circumference over 40 inches in a male or 35 inches in a female or BMI greater than 30.
3. Age between 18 and 70 years.
4. Stable on maximum tolerated dose of metformin for at least 3 months prior to enrollment.
5. Sedentary (less than 30 minutes per week of structured activity) and weight stable (2% body weight in past 6 months).
6. Metabolic syndrome based on NCEP ATP-3 guidelines with diabetes accepted as the glycemic component.
7. For women: at least 2 years postmenopausal, surgically sterile, or using an acceptable contraceptive regimen to include OCP, IUD, double barrier, depo-provera, or subcutaneous progestin implant and negative urine pregnancy test at trial start.
8. For men: surgically sterile or agreement that any female partner meet criteria of 7.

Exclusion Criteria:

1. Pregnancy, breast feeding, or planning to become pregnant during the study period.
2. GFR less than 60mL per minute per meter squared.
3. Any medical condition expected to be terminal within one year.
4. Cirrhosis of any cause or liver disease due to auto-immune, infectious or alcohol induced hepatitis.
5. Active mental illness or other condition which in the opinion of the investigator would prevent informed consent or compliance with study protocol.
6. Use of PPAR agonist within six months prior to enrollment.
7. Daily insulin use.
8. Allergy or intolerance of sitagliptin or other DPP-4 inhibitor.
9. Use of DPP-4 inhibitor, bile acid sequesterant, or weight loss medications within three months prior to enrollment.
10. Significant alcohol use defined as greater than 21 standard servings of alcohol (10gms) per week for men and greater than 14 for women.
11. History of bariatric surgery or planned bariatric surgery during the study period.
12. Weight, girth, or other factor preventing MRI scanning.
13. Receipt of another study drug within 30 days of screening.
14. Unable to receive a DEXA scan due to participating in research study or medical procedure involving ionizing radiation exposure equivalent to a chest x-ray or greater in the past 12 months.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-03; Primary Completion 2015-12 (Estimated); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Change in Liver steatosis | baseline and Six months
  Steatosis measured by Magnetic Resonance Spectroscopy

CONTACTS AND LOCATIONS:
Overall Officials: Michael Gardner, MD, Principal Investigator — University of Missouri-Columbia
Locations (1):
- University of Missouri-Columbia: Diabetes Center, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No